CLINICAL TRIAL: NCT07202585
Title: Analysis of Variability in the Management of Respiratory Infections in Hospitalized Patients Under 2 Years of Age Using Propensity Score Matching in Pediatric Inpatient Units"
Brief Title: Analysis of Variability in the Management of Respiratory Infections in Hospitalized Patients Under 2 Years of Age
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Principal Investigator, Juan Pablo Ferreira, Principal Investigator, Hospital General de Niños Pedro de Elizalde
Other Study IDs: Variability PMS
Record Dates: First submitted 2025-08-06; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Bronchiolitis; Bronchiolitis Acute Viral
Keywords: Acute Lower Respiratory Infections (ALRI); Pediatric Respiratory Infections; Clinical Variability; Propensity Score Matching
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Medical practice variability refers to differences in treatment and clinical outcomes that cannot be solely explained by patient characteristics or medical conditions. This variability can lead to inconsistent outcomes, especially in complex environments like pediatric inpatient wards. Standardization of care protocols is proposed as a way to reduce this inconsistency.

DETAILED DESCRIPTION:
Medical practice variability refers to differences in treatment and clinical outcomes that cannot be solely explained by patient characteristics or medical conditions. This variability can lead to inconsistent outcomes, especially in complex environments like pediatric inpatient wards. Standardization of care protocols is proposed as a way to reduce this inconsistency.

One key area of variability is the diagnosis and treatment of respiratory infections, particularly distinguishing bacterial from viral bronchial infections. Due to the lack of definitive clinical criteria, there is widespread antibiotic use (65-80% of cases), despite ongoing debate about their effectiveness.

Implementing standardized management protocols in pediatric wards aims to reduce such variability and improve clinical outcomes. This study will attempt to measure variability in outcomes based on treatment variables, identifying sources of medical variability and their impact.

ELIGIBILITY:
Inclusion Criteria:

Children under 2 years hospitalized with LARI in general pediatric wards during the winter months (June-September) of 2025 and 2026 in Buenos Aires

Exclusion Criteria:

Intensive care admission on entry Presence of comorbidities: congenital heart disease. Chronic respiratory conditions, neuromuscular diseases, immunodeficiencies,.

Prolonged previous hospitalizations for unrelated causes Severe disabilities influencing hospitalization duration.

Ages: 1 Month to 24 Months | Sex: All
Age Groups: Child
Study Population: Children under 2 years hospitalized with LARI in general pediatric wards during the winter months (June-September) of 2025 and 2026 in Buenos Aires
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Variability in the treatment:Length of Hospital Stay | 2 years
  * Definition: Total number of full calendar days from admission to pediatric ward until medical discharge.
  * Measurement: Recorded in patient's medical record. Calculated as discharge date - admission date.
  * Type of Variable: Continuous (days).
  * Analysis: Mean/median days compared between groups after Propensity Score Matching.

SECONDARY OUTCOMES:
Explore Clinical outcomes | 2 years
  * Definition: Incidence of adverse events during hospitalization, including nosocomial infections, escalation to ICU, or other significant medical complications.
  * Measurement: Categorical (Yes/No for each complication) documented in medical record with onset and resolution dates.
  * Type of Variable: Binary for each event; total count of events per patient can also be analyzed.
  * Analysis: Proportion of patients experiencing ≥1 complication compared between groups after Propensity Score Matching.

CONTACTS AND LOCATIONS:
Locations (1):
- HGNPE, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
all data will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years

REFERENCES:
- [Background] Kane LT, Fang T, Galetta MS, Goyal DKC, Nicholson KJ, Kepler CK, Vaccaro AR, Schroeder GD. Propensity Score Matching: A Statistical Method. Clin Spine Surg. 2020 Apr;33(3):120-122. doi: 10.1097/BSD.0000000000000932. PMID 31913173